CLINICAL TRIAL: NCT04246645
Title: Effect of Core Stability Exercises on Hand Functions in Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: hanaa mohsen (Other)
Responsible Party: Sponsor-Investigator, hanaa mohsen, lecturer in the deparment of pediatrics and peditaric surgery , faculty of phyical therapy, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hana 2
Record Dates: First submitted 2020-01-21; First posted 2020-01-29 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): received the selective physiotherapy exercises
- STUDY GROUP (Experimental): received the same selective physiotherapy exercises program in addition to core stability exercises three times/week for 60 min for 12 weeks
  Interventions: Other: CORE STABILITY EXERCISES

INTERVENTIONS:
Other: CORE STABILITY EXERCISES — SELECTED CORE EXERCISES
  Arms: STUDY GROUP

SUMMARY:
Background: Impaired upper extremity is the major disability facing the children with hemiplegia as the inability to use hands for reach; grasp and manipulation affect their daily life activities. little attention has been given to gain perspective about abnormal movements that are detectable in hemiplegic cerebral palsy that are related to one's level of core stability and how they affect their hand functions.

DETAILED DESCRIPTION:
Background: Impaired upper extremity is the major disability facing the children with hemiplegia as the inability to use hands for reach; grasp and manipulation affect their daily life activities. little attention has been given to gain perspective about abnormal movements that are detectable in hemiplegic cerebral palsy that are related to one's level of core stability and how they affect their hand functions.

Objective: The purpose was to investigate the effectivness of core stability exercises on hand functions in hemiplegic cerebral palsy.

Methods: Thirty hemiparetic cerebral palsied children of both sexes, ranged in age from 6 to 8 years enrolled in this study. They randomly assigned into two groups of equal number. Group (A) received the selective physiotherapy exercises and group (B) received the same selective physiotherapy exercises program in addition to core stability exercises three times/week for 60 min for 12 weeks. Time motor performance, gross manual dexterity and skills of the upper extremity were assessed by using Jebsen Taylor Test (JTHFT), Box and Block Test (BBT) and Quality Upper Extremity Skill Test (QUEST) respectively before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The level of gross motor function ranged from II to III, according to Gross Motor Function Classification System
* All participants are cognitively capable and competent of interpreting and following instructions

Exclusion Criteria:

* if they had fixed contractures or deformities of the spine, upper or lower extremities,
* visual or respiratory disorders, orthopedic surgery on their involved upper extremity;
* dorsal rhizotomy;
* botulinum toxin therapy in the upper extremity musculature during the past 6 months
* who wished to receive it within the period of study

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor Test | Jebsen Taylor Test used to assess gross manual dexterity before the intervention and after three months of the intervention . the loweest score indicate improvement
  scale used to asses gross manual dexterity

SECONDARY OUTCOMES:
Box and Block Test | Box and Block Test used to asses gross manual dexterity pre and after 3 months of intervension
  scale used to asses gross manual dexterity
Quality Upper Extremity Skill Test | Quality Upper Extremity Skill Test scale used to asses skills of the upper extremity pre and after 3 months of intervension
  scale used to asses skills of the upper extremity

CONTACTS AND LOCATIONS:
Locations (1):
- Badr Univesity in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No